CLINICAL TRIAL: NCT05149703
Title: Efficacy of Postural Reeducation in Elite Gymnasts With Back Pain. A Randomized Clinical Trial
Brief Title: Efficacy of Postural Reeducation in Elite Gymnasts With Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Juan Martínez Fuentes, Study Director, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE102105
Record Dates: First submitted 2021-11-19; First posted 2021-12-08 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Back Pain; Back Strain Lower Back; Athletic Injuries
Keywords: Physiotherapy; Rehabilitation; Treatment; Isostretching; Postural treatment
MeSH Terms: conditions — Back Pain; Athletic Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mezieres Group (Experimental): This intervention includes a total of three postures of the Mézières therapy. Specifically, the postures maintained for 12 weeks consist of: supine dancer; in supine position with the upper extremities abducted 120 °; and dancer in a sitting position.
  Interventions: Other: Mezieres Postural Treatment
- Isostretching Group (Active Comparator): This study aims to follow a total of 6 isostretching postures, the most similar to the Mezieres method. In each of the isostretching positions, if it is symmetric, 3, 6 or 9 repetitions will be performed and if it is asymmetric, 2, 4, or 8 repetitions.
  Interventions: Other: Mezieres Postural Treatment

INTERVENTIONS:
Other: Mezieres Postural Treatment — Implementation of 12 weeks suitable postures of Mezieres method

SUMMARY:
Introduction: Low back pain is a musculoskeletal disorder that is associated with symptoms such as pain, limitation of joint range and postural problems in athletes. Methods: The study design is a randomized controlled clinical trial with a minimum of 35 elite gymnasts with back pain. Two postural treatments will be implemented, Mezieres Method and Isostretching to verify if there is improvement of back pain in gymnasts and to compare both procedures. Discussion: This trial could generate a greater understanding of the importance of posture related to low back pain and its possible treatments.

DETAILED DESCRIPTION:
A randomized controlled clinical trial with two groups (intervention and placebo) will be implemented. The intervention group will have the Mezieres technique as postural treatment while the placebo group will follow a total of 6 isostretching positions.

In total, the two treatments with 30 minutes and duration or with a frequency of 2 weekly sessions will be implemented for a period of 12 weeks. All treatments will be performed by the same certified therapist and with a minimum of 5 years of experience in postural treatments. The measurements will be made immediately after the first session, in 2 weeks, 6 weeks and in the last week of intervention by a blind researcher who did not participate in the treatments, but with experience in this field.

ELIGIBILITY:
Inclusion Criteria:

* Elite gymnastic athletes with low back pain
* Active participation in the national competition
* Practice at least three times a week for 60 minutes
* Minimum training time of 7 hours a week

Exclusion Criteria:

* Gymnast whom suffer from chronic disease or acute musculoskeletal injury
* Herniated disc
* Spondylolisthesis

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Back status | 12 weeks
  Measured with Oswestry questionaire. It consists of 10 categories. Each category consists of 6 items scored from 0 to 5 with the first statement scoring 0 until the last statement scoring 5.
Back disability | 12 weeks
  Measured with Roland Morris Questionaire wich consist in 24 points of back disability actual phrases
Range of motion | 12 weeks
  Measured with Baiobit software
Pain intensity | 12 weeks
  Measured with Numeric Rating Scale wich consist in measure pain intensity with a score of 0-10

SECONDARY OUTCOMES:
Subjetive tension perception | 12 weeks
  Measured with Borg Scale, which include a rating of 6 perceiving "no exertion at all" to 20 perceiving a "maximal exertion" of effort.
Spinal curvature evaluation | 12 weeks
  Measured with Spinal Mouse Software
Stiffness test | 12 weeks
  Measured with Baiobit software
Posture stability | 12 weeks
  Measured with stabilometry with a duration of 50 seconds with Lizard posturometric and stabilometric platform

CONTACTS AND LOCATIONS:
Overall Officials: Juan Martínez Fuentes, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Universidad Católica de Murcia, Murcia, Spain